CLINICAL TRIAL: NCT06148961
Title: Effect of Botox Before Modified Lip Repositioning and Modified Lip Repositioning Only in Relapse of the Excessive Gingival Display Within One Year
Brief Title: Effect of Botox Before Modified Lip Repositioning Repositioning Only in Relapse of the Excessive Gingival Display Within One Year
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Cherine Emad Mahmoud Mohamed Hamada, assistant lecturer, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-2025
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Excessive Gingival Display

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): botox injection prior to surgical intervention by 5 to 10 days A surgical marker was used to outline the boundaries of the surgical incision region.
  the height of the superior incision was measured as 15 mm within the vestibule. Superior and inferior incisions were made with a scalpel blade number 15 and linked bilaterally by two vertical incisions.
  A partial thickness dissection was used to remove the strip of the indicated mucosa, exposing the fascia of the connective tissue beneath. When necessary, all salivary glands and frenal attachments were removed. The surgical site was then properly closed using a periosteal simple interrupted suture was put in place prior to the continuous interlocking sutures. It was placed by commencing the needle 2 mm coronal to Per surgery site, 3 to 4 periosteal sutures were typically The new mucosal boundary to the gingiva was stabilized in its new place using this suture
  Interventions: Procedure: botox prior to modified lip repostioning
- control group (Active Comparator): A surgical marker was used to outline the boundaries of the surgical incision region.
  the height of the superior incision was measured as 15 mm within the vestibule. Superior and inferior incisions were made with a scalpel blade number 15 and linked bilaterally by two vertical incisions.
  A partial thickness dissection was used to remove the strip of the indicated mucosa, exposing the fascia of the connective tissue beneath. When necessary, all salivary glands and frenal attachments were removed. The surgical site was then properly closed using a periosteal simple interrupted suture was put in place prior to the continuous interlocking sutures. It was placed by commencing the needle 2 mm coronal to Per surgery site, 3 to 4 periosteal sutures were typically The new mucosal boundary to the gingiva was stabilized in its new place using this suture
  Interventions: Procedure: botox prior to modified lip repostioning

INTERVENTIONS:
Procedure: botox prior to modified lip repostioning — botox injection prior to surgical intervention by 5 to 10 days A surgical marker was used to outline the boundaries of the surgical incision region.
  the height of the superior incision was measured as 15 mm within the vestibule. Superior and inferior incisions were made with a scalpel blade number 15 and linked bilaterally by two vertical incisions.
  A partial thickness dissection was used to remove the strip of the indicated mucosa, exposing the fascia of the connective tissue beneath. When necessary, all salivary glands and frenal attachments were removed. The surgical site was then properly closed using a periosteal simple interrupted suture was put in place prior to the continuous interlocking sutures. It was placed by commencing the needle 2 mm coronal to Per surgery site, 3 to 4 periosteal sutures were typically The new mucosal boundary to the gingiva was stabilized in its new place using this suture

SUMMARY:
The growing interest of patients in esthetic procedures, as well as the development of less invasive protocols in dentistry, has promoted the development of treatment plans that include stability, harmony, and function in orofacial rehabilitation.

Poor esthetics interfere with an individual's personal, social, and professional relationships and is an individual consideration that varies according to the patient's age, time, region, and culture concerning what is considered beautiful.

DETAILED DESCRIPTION:
People are increasingly being inspired to get more corrective and cosmetic surgeries as an esthetic smile becomes a more fundamental component of what it means to be beautiful.

There are several variables that affect how appealing and esthetic a smile is Esthetic perception varies according to cultural, societal, environmental, and individual factors like experience and educational level Previous studies have shown that a smile with less gingival display (GD) is viewed as more beautiful, with dental professionals being more critical of gingival presentation than laypeople According to research by several authors, the ideal GD ranges from 1 to 3 mm While many factors influence how pleasant a smile is seen, excessive GD (EGD), sometimes referred to as a gummy smile, is regarded as a key factor in smile analysis and one of the main issues connected to an unsatisfactory dental smile.

To reduce the relapse associated with repositioning surgery and to provide a lasting treatment without the need for reapplication, as in the case of the toxin, a combined treatment using the toxin preoperatively was considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients that is not satisfied with his smile having excessive gingival display
* Adult Age ≥ 21 years.
* Systemically and periodontally Healthy patients.
* had gingival exposure greater than 3 mm when smiling
* had a hyperactive upper lip with or without other causes of EGD (lip displacement ≥ 9 mm) before botox & ≥ 3mm after.
* Cooperative patients able and accept to come for follow up appointments.

Exclusion Criteria:

* • smoking

  * pregnancy or lactation
  * Systemic diseases; neuromuscular,neurological, or psychological disorders or consumption of controlled medication
  * Patients having medical condition or any drugs that could affect healing
  * Patients with systemic condition that can't undergo minor oral surgery
  * Patient allergic to Botox or multiple allergic conditions
  * have history of previous Botox injection
  * periodontal disease
  * excessive gingival display at rest
  * those who declined the informed consent or who did not consent to the risks described.
  * Those who have deviate smile

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in gingival display | 3,6&12 months
  Using a 15-cm marked ruler (Antunes et al., 2022)

SECONDARY OUTCOMES:
Patient's satisfaction | 3,6 &12 months
  Survey (Silva et al., 2013)

OTHER OUTCOMES:
Maintenance of reduction of gingival display | 3 , 6 & 12 months
  callipper

CONTACTS AND LOCATIONS:
Locations (1):
- Cherine Emad Mahmoud Mohamed Hamada, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided